CLINICAL TRIAL: NCT01631877
Title: Efficacy and Safety of Acenocoumarol for Treatment of Nontumor Portal Vein Thrombosis in Cirrhosis of Liver
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS- PVT-01
Record Dates: First submitted 2012-06-15; First posted 2012-06-29 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-12

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Enoxaparin; Acenocoumarol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- enoxaparin with acenocoumarol (Experimental): Patients will receive enoxaparin 100mcg/kg for 5days along with acenocoumarol 2mg with titration of dose to maintain a target INR of 2-3.intially the INR will be monitored twice weekly with gradual escalation of dose to achieve target INR.After achieving the target INR this is to be repeated every 4th weekly. The Doppler Ultra Sonography screening will be done every 3monthly to assess the recanalization of portal vein thrombus but the medications will be continue for one year irrespective of recanalization.
  Interventions: Drug: Enoxaparin with acenocoumarol
- Placebo (Placebo Comparator): Injection placebo will be given for 5 days along with placebo tablets.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Enoxaparin with acenocoumarol — enoxaparin 100mcg/kg for 5days along with acenocoumarol 2mg to start with and dose to be adjusted for the target INR
  Arms: enoxaparin with acenocoumarol
Other: placebo — injection placebo will be given for 5 days along with placebo tablets
  Arms: Placebo

SUMMARY:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have non tumor portal vein thrombosis will be enrolled. The baseline Doppler parameter will be recorded and the patient will be randomized into either interventional (acenocoumarol) or placebo group along with first five days of subcutaneous Low Molecular Weight Heparin inj. Enoxaparin in the interventional arm and placebo injection in the control arm. Every 3 monthly the Doppler screening for recanalization of portal vein thrombus will be done with monitoring of International Normalized Ratio (INR)with target INR 2-3. Both the groups will receive the therapy for one year irrespective of the Doppler findings in relation to portal vein thrombus re-canalization.Then one year drug free monitoring will be done in both the groups as per the primary or secondary outcome. .

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis
* Partial or total Portal vein thrombus (evidence of chronic thrombus)
* Informed consent to participate in the study

Exclusion Criteria:

* Acute thrombus in Portal vein
* Hepatocellular carcinoma or any other malignancy,
* Hypercoagulable state other than the liver disease related
* DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs.
* Base line INR >2
* Child Turcott Pugh score>11
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy.
* Uncontrolled Hypertension
* Age>70 yrs
* Non responders to beta-blocker requiring Endoscopic Variceal Ligation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Proportions of patients who will achieve Recanalization of thrombus (complete i.e No thrombus is seen or partial i.e up to 50% of the lumen become patent.)on oral anticoagulant acenocoumarol during the study period of 2 year from randomization. | 2 years

SECONDARY OUTCOMES:
Proportions of patients who will show improvement in Child Turcott Pugh (CTP) (>2 points)in both groups | 2 years
Proportions of patients who will show improvement in Model for End Stage Liver Disease (MELD)(>4 points)in both groups | 2 years
Proportions of patients who will achieve reduction in liver stiffness > 5 Kpa by transient elastography in both groups | 2 years
Proportions of patients will show decrease in hepatic decompensation i.e hepatic encephalopathy,ascites,hepato renal syndrome,variceal bleed,jaundice and coagulopathy in both groups. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences., New Delhi, National Capital Territory of Delhi, India